CLINICAL TRIAL: NCT06832995
Title: Incidence and Risk Factors for Post-Anesthetic Morphine Titration in Recovery Room After Hip and Knee Arthroplasties: a Single-center Retrospective Study
Brief Title: Incidence and Risk Factors for Post-Anesthetic Morphine Titration in Recovery Room After Hip and Knee Arthroplasties
Acronym: PAMTA
Status: Active, not recruiting | Type: Observational
Sponsor: Hôpital Privé Sévigné (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-HPS
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Arthropathy of Hip; Arthropathy of Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group T: IV morphine administered during the PACU stay
  Interventions: Drug: IV morphine administered during the PACU stay
- group NT: no titration required in PACU

INTERVENTIONS:
Drug: IV morphine administered during the PACU stay — IV morphine administered during the PACU stay
  Groups: group T: IV morphine administered during the PACU stay

SUMMARY:
Despite the use of multimodal analgesia combining nerve block (NB) and systemic analgesia, intravenous (IV) morphine titration in the post-anesthetic care unit (PACU) after total hip (THA) and knee (TKA) arthroplasty is required to relieve early moderate-to-severe pain. Sedation occurrence during titration and a VAS score higher than 60/100mm are two independent risk factors for postoperative pain during hospitalization.

The association of NB and multimodal analgesia constitutes the reference in evidence-based recommendations. An adductor or femoral triangle block, alone or associated with periarticular infiltration, is recommended during TKA. During THA, NB associated with surgical periarticular infiltration improves analgesia and rehabilitation This study aims to identify the incidence and risk factors of morphine titration in PACU after lower limb arthroplasty performed by 5 experienced surgeons and using a multimodal analgesic procedure

ELIGIBILITY:
Inclusion Criteria:

* Total hip arthroplasty
* Total Knee Arthroplasty
* Uni-compartmental knee arthroplasty (UKA)

Exclusion Criteria:

* Bilateral surgery Surgical revision Hip fracture surgery Other osteoarticular procedure(s) associated to hip/knee arthroplasty Refusal to use data Contra-indication of paracetamol, ketoprofen and dexamethasone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each patient who underwent unilateral knee, total knee and total hip arthroplasty at the Sévigné Private Hospital between January 1, 2023, and December 31, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
morphine titration | after surgery, in the post-anesthetic care unit

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Sévigné, Cesson-Sévigné, France

IPD SHARING:
Plan to Share IPD: No